CLINICAL TRIAL: NCT04692428
Title: Fracture of the Upper Femoral Extremity in the Elderly Patients: Comparison of the Supra-inguinal Fascia Iliaca Block VS Femoral Nerve Block Ultrasound Guided in the Positioning and Post-operative Analgesia for Spinal Anesthesia
Brief Title: Comparison of the Ultrasound Supra-inguinal Fascia Iliaca Block vs Femoral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Mechaal Benali, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UTEM FIBSI
Record Dates: First submitted 2020-12-25; First posted 2020-12-31 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Hip Fracture
Keywords: analgesia; hip fracture; nerve block
MeSH Terms: conditions — Hip Fractures; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIBSI group (Experimental): ultrasound supra inguinal Fascia iliaca block
  Interventions: Procedure: Locoregional analgesia
- FNB group (Experimental): ultrasound femoral nerve block
  Interventions: Procedure: Locoregional analgesia

INTERVENTIONS:
Procedure: Locoregional analgesia — the supra-inguinal fascia iliaca block versus the femoral nerve block

SUMMARY:
Patients were randomly assigned to tow groups: infrainguinal ultrasound guided iliaca fascia block (FIBSI) and femoral nerve block (FNB) for FIBSI, the probe is placed transversely between anterior superior iliac spine (ASIS) and the pubic spine. The transducer is translated laterally to identify the Sartorius muscle. Cephalic inclination of the probe. The medial end of the transducer faces towards the umbilicus, which is the final position. The 100mm neurostimulation needle is advanced in the In Plan approach to pass through the iliac fascia. Once the correct position is confirmed, 30 ml of 1% Ropivacaine is gradually injected between the iliac fascia and the iliac muscle.

For FNB, the probe was placed under the inguinal ligament. The femoral vessels and the nerve section are visualized; The 100mm neurostimulation needle is advanced in the In Plan approach and 30ml of 1% Ropivacaine has been injected along the nerve sheath

DETAILED DESCRIPTION:
Patients were randomly assigned to tow groups: infrainguinal ultrasound guided iliaca fascia block (FIBSI) and femoral nerve block (FNB) for FIBSI,the probe is placed transversely between the EIAS and the pubic spine,The transducer is translated laterally to identify the sartorius muscle. Cephalic inclination of the probe: The iliac muscle is located at the medial border in the shadow of the superior anterior iliac spine.The medial end of the transducer faces towards the umbilicus, which is the final position.

The anatomy identified, from superficial to deep, consisting of subcutaneous fat, internal oblique muscle, transverse abdominal muscle, iliaca fascia covering the iliac muscle. The 100mm neurostimulation needle is advanced in In Plan approach to cross the iliaca fascia. With the tip of the needle just below the iliaca fascia, 2 ml of local anesthetic was injected to confirm the location of the tip. Once the correct position is confirmed, 30 ml of 1% Ropivacaine is gradually injected between the iliac fascia and the iliac muscle.

for FNB,The probe was placed under the inguinal ligament. Femoral vessels and sectional nerve are visualized. The nerve was located, an 100mm neurostimulation needle is advanced in In Plan approach, and 30 ml of 1% Ropivacaine was injected along the nerve sheath.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) class I, II, and III patients scheduled for emergency surgery with the diagnosis of proximal femur fracture

Exclusion Criteria:

* hemorrhagic diathesis,
* peripheral neuropathies,
* allergy to amide local anaesthetics,
* mental disorders,
* those on analgesics within 8 hour prior to performing nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Positioning pain before performing spinal anesthesia | 20 minutes after realization of blocks
  Pain in positioning was assessed by measuring the simple verbal scale (0= no pain- 4= worst pain possible) after 20 minutes for realization block

SECONDARY OUTCOMES:
Postoperative pain | at the third, sixth, twelfth and twenty-four hours postoperatively
  Postoperative pain was assessed by the Simple Verbal Scale (SVS) at the third, sixth, twelfth and twenty-four hours postoperatively
quality of patient placement in the sitting position | after 20 minutes of realization of block
  The quality of patient positioning was subjectively rated as unsatisfactory, good or optimal depending on the ease of positioning for spinal anesthesia
The level of sensory block at 20 minutes after realization of block | before and 20 minutes after realization of blocks
  The quality of the sensory block was evaluated by the PinPrick Test in the external, internal and anterior part of the thigh in comparison with the same stimulation at the level of the contralateral limb.
  using a sterile needle at 20 minutes after realization of block on the territory of femoral, obturator and lateral cutaneous nerve of the thigh
Patient satisfaction | five minutes after the end of the realization of spinal anesthesia
  Patient satisfaction was evaluated after completion of spinal anesthesia by using a two-point score: 1= good, if necessary, I'll repeat it and 2= bad, I will never repeat it again.

CONTACTS AND LOCATIONS:
Overall Officials: mechaal benali, PROFESSOR, Principal Investigator — university manar Tunis tunisia
Locations (1):
- Mechaal Benali, Nabeul, Mrezga, Tunisia